CLINICAL TRIAL: NCT07349797
Title: An Open Label, Single-Center, Safety and Pharmacokinetic Study of Lumitrace® Injection (Relmapirazin) and the Use of the MediBeacon® Transdermal GFR System Using the TGFR Reusable Sensor With TGFR Disposable Ring for the Evaluation of Kidney Function in Patients With Heart Failure
Brief Title: MediBeacon® Transdermal GFR System for the Evaluation of Kidney Function in Adults With Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 100-300
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Glomerular Filtration Rate; Heart Failure
Keywords: Relmapirazin; Lumitrace
MeSH Terms: conditions — Heart Failure | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 130 mg Lumitrace/1.5 mL Iohexol (Experimental): Participants will have the tGFR sensor placed and background measurements initiated. Participants will then receive a single intravenous 130 mg dose of Lumitrace followed by 1.5 mL of iohexol. They will be followed at the study center for 10-24 hours.
  Interventions: Device: Lumitrace; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (tGFR); Drug: Iohexol

INTERVENTIONS:
Device: Lumitrace — 18.6 mg/mL in a 7.0 mL volume administered by intravenous injection over 30 - 60 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 - 60 seconds
  Other Names: Relmapirazin
Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (tGFR) — Site staff will place and affix the tGFR reusable sensor and Disposable Ring for all enrolled participants. One sensor will be attached to the upper chest. An adhesive clip, surgical tape or other means may also be used to alleviate tension on the sensor cord. TGFR assessments will be collected for a minimum of 6 hours up to 8 hours post Lumitrace injection.
Drug: Iohexol — 1.5 mL of a 647 mg/mL solution administered by intravenous injection over 30 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 -60 seconds
  Other Names: Omnipaque 300

SUMMARY:
The goal of this clinical trial is to evaluate the accuracy and feasibility of transdermal glomerular filtration rate (tGFR) assessment using relmapirazin (Lumitrace) and the MediBeacon tGFR system compared to plasma clearance measurement of GFR in adults with heart failure.

The main question it aims to answer is the comparison of the transdermal-derived GFR for each participant using the MediBeacon tGFR to their nGFRBSA measurement.

Participants will participate in a Screening visit that will take place within 15 days of the scheduled administration of Lumitrace and iohexol. On dosing day, participants will have the tGFR reusable sensor with disposable adhesive ring placed on their chest, and the MediBeacon Transdermal GFR System initiated to collect background fluorescence. Following an injection of Lumitrace and iohexol and the initiation of GFR assessments, participants will be followed at the study center for 10-24 hours. All participants will participate in a follow-up phone call approximately 7 days after the last exposure to Lumitrace and iohexol. Researchers will analyze the results to compare the tGFR values to the nGFRBSA measurements for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;

   1. Eligible female non-pregnant participants who are either not of child-bearing potential or willing to use adequate contraception during the trial
   2. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post-dose
   3. For women of child-bearing potential, the participant should have a negative serum pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization
   4. Men will not donate sperm during the study and for 1 month following the last dose of study drug.
2. Diagnosis of symptomatic heart failure: Subject has symptomatic heart failure, ACC/AHA Stage C or D, ambulatory or hospitalized for heart failure, adjudicated by a principal investigator, and meeting both of the following:

   1. Clinical syndrome: Symptoms and/or signs consistent with heart failure (e.g., dyspnea, fatigue, edema, rales, elevated JVP), and
   2. Objective evidence of heart failure (≥1 of):

      * Left ventricular systolic dysfunction or other structural abnormalities (left atrial enlargement, left ventricular hypertrophy, diastolic dysfunction on echocardiography) or
      * Hemodynamic evidence of elevated filling pressures by invasive or noninvasive assessment, or
      * Elevated natriuretic peptides obtained within 90 days from enrollment: NT-proBNP ≥300 pg/mL (BNP ≥100 pg/mL) in sinus rhythm or NT-proBNP ≥900 pg/mL (BNP ≥300 pg/mL) in atrial fibrillation
3. Participants who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
4. Adequate venous access sufficient to allow blood sampling per protocol requirements

Exclusion Criteria:

To be eligible for the study, participants must not meet any of the criteria noted below:

1. Intolerance to iohexol or iodine allergy
2. Known allergy to relmapirazin or severe hypersensitivity reactions to adhesives or related products
3. Administration of iohexol for cross-sectional imaging within a week from the dosing visit
4. Limb amputation
5. Primary kidney disease (e.g., glomerulonephritis or polycystic kidney disease)
6. Acute kidney injury (AKI) or unstable kidney function at the time of dosing visit
7. Clinical signs of excessive volume overload (edema grade 3-4 or ascites)
8. Significant scarring, tattoos, or alterations in pigmentation on the sternum or other sensor location areas that would alter sensor readings
9. Use of tanning sprays, tanning products, etc. on the upper chest within 2 weeks of dosing day
10. Use of make-up, lotions, Vaseline or other products on the area of the upper chest on the day prior to or the day of dosing
11. Participants who have received nephrotoxic agent or signs or symptoms suggestive of a condition that may result in acute kidney injury within two weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of Transdermal Derived Glomerular Filtration Rate (tGFR) to the Plasma-derived Indexed Glomerular Filtration Rate (nGFR) | Day 1
  The performance measure of P30 is defined as the proportion of transdermal derived GFR values that are within 30% of the measured plasma-derived GFR across all participants. The comparison of transdermal derived glomerular filtration rate (tGFR) with respect to the plasma-derived indexed glomerular filtration rate (nGFR) will be calculated with a double-sided 95% confidence interval (CI). The performance goal is 0.75, and success for the study is defined as a lower limit of the 95% CI greater than 0.75.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon, Inc.
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No